CLINICAL TRIAL: NCT01014429
Title: A Phase I Dose Escalation Study of NMS-1286937 Administered to Adult Patients With Advanced/Metastatic Solid Tumors
Brief Title: Study of NMS-1286937 in Adult Patients With Advanced/Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLKA-937-001
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Phase I dose escalation study; Advanced or metastatic solid tumors; PLK 1 inhibitor; Adult patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: NMS-1286937

INTERVENTIONS:
Drug: NMS-1286937 — Single Arm, dose escalation study. No. of cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of NMS-1286937, a polo-like-kinase 1 inhibitor, in patients with advanced metastatic solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/metastatic solid tumors, for which no effective standard therapy exist
* Adult patients (age >/= 18)
* ECOG performance status (PS) 0 or 1
* Life expectancy of at least 3 months
* Adequate renal, liver function and bone marrow reserve
* Prior cancer therapy allowed, with max 4 regimens of chemotherapy. Washout: at least 4 wks (6 wks for nitrosoureas, mitomycin C and liposomal doxorubicin) and all toxicities recovered to CTC Grade </=1
* Prior radiotherapy allowed if no more than 25% of BM reserve irradiated
* Women and men of child producing potential should agree to use effective contraception
* Capability to swallow capsules intact

Exclusion Criteria:

* Known uncontrolled/symptomatic brain metastases
* Currently active second malignancy
* Major surgery in the last 4 wks
* Any of the following in the past 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis
* Pregnancy or breast-feeding women
* Known active infections
* History of drug allergic reactions
* Gastrointestinal disease or other malabsorption syndromes that would impact on drug absorption.
* Documented gastrointestinal ulcer
* Other severe concurrent acute or chronic medical or psychiatric condition that could compromise protocol objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and first cycle dose limiting toxicities (DLTs) | Cycle 1

SECONDARY OUTCOMES:
Evaluation of pharmacokinetics: plasma concentration at different times after dosing, area under the curve (AUC), maximum plasma concentration (Cmax), clearance (CL), volume of distribution, half-life (t½) | Cycles 1 and 2
Evaluation of pharmacodynamics: biomarkers modulation in skin and/or tumor samples of consenting patients | Cycles 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Mariani, Biol Sci D, Study Director — Nerviano Medical Sciences; Maria Adele Pacciarini, Biol Sci D, Study Director — Nerviano Medical Sciences; Glen J Weiss, MD, Principal Investigator — Arizona TGen Clinical Reserch Services at Scottsdale Healthcare
Locations (1):
- Arizona TGen Clinical Research Services at Scottsdale Heathcare, Scottsdale, Arizona, United States